CLINICAL TRIAL: NCT07191561
Title: Mechanisms in Hepatic Lipid Metabolism in Alcohol Use Disorder: From Genomics, Transcriptomics to Metabolomics
Brief Title: Hepatic Lipid Metabolism-Alcohol Use Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001764; 001764-DK
Record Dates: First submitted 2025-09-24; First posted 2025-09-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-22

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Liver; Biopsy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver biopsy: All participants in the study will undergo liver biopsies
  Interventions: Diagnostic Test: Liver biopsy

INTERVENTIONS:
Diagnostic Test: Liver biopsy — Biopsy of the liver

SUMMARY:
Patients with hepatic steatosis due to alcohol will be offered liver biopsies when they enter a detoxification program. The first biopsy will occur in the first week of admission and the second in the fourth week when the steatosis has resolved. The hepatic transcriptome will be compared,

DETAILED DESCRIPTION:
Study Description:

The liver is central to lipid metabolism, intimately involved with lipid uptake, lipoprotein synthesis and lipid synthesis. Alcohol has known effects on changing lipid composition including increases in HDL and decreases in LDL; nevertheless, the underlying mechanisms of this altered lipoprotein metabolism is not understood. Current spectroscopy data characterize the changes in lipoprotein profiles with alcohol cessation. We aim to study liver lipid metabolism by performing liver biopsies and transcriptome analysis in participants with alcohol use disorder.

Objectives:

Primary Objective:

To understand the transcriptomics of hepatic lipid metabolism in alcohol use disorder

Secondary Objective:

To understand other transcriptome changes in alcohol use cessation.

Tertiary Objective:

To elucidate the genomics-transcriptomics-metabolomics pathway of hepatic lipid metabolism in alcohol use disorder.

Endpoints:

Primary Endpoints:

-Transcriptome changes in lipid metabolism between week 1 and week 4.

Secondary Endpoints:

-Other transcriptome changes between week 1 and week 4.

Tertiary Endpoints:

* To make connections with existing genetics and metabolomics data with transcriptomics.
* Stool microbiome studies

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Any individual >=18 years of age who is enrolled in 14-AA-0181 and is seeking inpatient treatment.
* Vibration Controlled Elastography parameters with initial CAP of >295dB/m.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy
* Existing diagnosis of hyperlipidemia or essential hypertension
* Hemoglobin A1c >= 6.5%
* Waist to hip ratio: >=0.90 in males, >=0.85 in females
* Existing use of cholesterol lowering medications including statins, fibrates, or other similar medications used for the purposes of treating hyperlipidemia.
* Those with evidence of severe alcoholic hepatitis with a Maddrey s Discriminant Function > 32
* Those with other chronic liver diseases including chronic hepatitis B (positive hepatitis B surface Ag on admission), hepatitis C (positive hepatitis C RNA), or autoimmune hepatitis (clinical diagnosis based on high titer of positive ANA and or anti smooth muscle Ab and a history of autoimmune disease)
* HIV infection
* Contraindication or inability to perform a liver biopsy.

  * Participants with coagulopathy (PT/PTT values that are prolonged (Bullet) 3 seconds from the upper limit of the normal, including treatment with oral and parenteral anticoagulants), thrombocytopenia (< 70,000), abnormal bleeding time or platelet dysfunction. Antiplatelet agents taken for cardiovascular prevention will not exclude participants, unless they cannot be stopped safely for the performance of a liver biopsy.
  * Hemoglobin level < 11 g/dL
  * Inability to provide informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with alcohol use disorder, currently under inpatient treatment at the NIH.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Transcriptome changes in lipid metabolism between week 1 and week 4 of alcohol cessation. | November 2029
  Analysis of liver biopsies

SECONDARY OUTCOMES:
Other transcriptome changes between week 1 and week 4 of alcohol cessation | November 2029

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001764-DK.html